CLINICAL TRIAL: NCT06040476
Title: A Phase II, Randomized, Double-blind, Parallel, Placebo-controlled Study to Assess the Safety and Efficacy of Human Umbilical Cord Blood Infusion in Patients with Acute Ischemic Stroke
Brief Title: Human Umbilical Cord Blood Infusion in Patients with Acute Ischemic Stroke (AIS)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: StemCyte, Inc. (Industry)
Collaborators: StemCyte Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: StemCyte International, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCAS001
Record Dates: First submitted 2023-08-31; First posted 2023-09-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group: hUCB treatment (Experimental): Human cord blood infusion
  Interventions: Biological: hUCB
- B group: Placebo treatment (No Intervention): Placebo infusion

INTERVENTIONS:
Biological: hUCB — hUCB
  Arms: A group: hUCB treatment

SUMMARY:
A Phase II, Randomized, Double-blind, Parallel, Placebo-controlled Study to Assess the Safety and Efficacy of Human Umbilical Cord Blood Infusion in Patients with Acute Ischemic Stroke

DETAILED DESCRIPTION:
This is a phase II study to evaluate the safety and efficacy in hUCB treatment on the patients with acute ischemic stroke (AIS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥18 and ≤80 years of age.
* Subject with a confirmed diagnosis of AIS and hemiplegia

Exclusion Criteria:

* Subject with known immune disease, immunodeficiency, or receives immunosuppressive therapy/immunomodulators within 4 weeks or 5 half-lives prior to screening, whichever is longer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
safety-TEAE | From screening to 48 weeks
  Frequency and incidence of treatment-emergent adverse events (TEAEs).

IPD SHARING:
Plan to Share IPD: No